CLINICAL TRIAL: NCT04092504
Title: Optimized Recovery After Trauma in Geriatric Patient (Gero - ERAT)
Brief Title: Optimized Recovery After Trauma in Geriatric Patient
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 766-18
Record Dates: First submitted 2019-05-29; First posted 2019-09-17 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Geriatric Assessment; Quality of Life; Trauma; Fragility; Injury; Rehabilitation; Recovery
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Implementation research with control group
Who Masked: Participant
Masking Description: Elderly trauma patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard care at the unit
- Gero-Erat (Experimental): New care pathway that is built on the concept of ERAS and CGA
  Interventions: Other: gero-erat

INTERVENTIONS:
Other: gero-erat — The intervention is a standardize Care Plan which will be developed based on the evidence of caring for elderly patients in a trauma setting. The Care Plan will have its base in, the concept of ERAS and CGA. Also, patient experience will be taken in consideration and complement the care pathway.
  Patients admitted to the trauma unit will be given the care and asked to be a part of the study witch include to fill out surveys at baseline, six months and 1 year.
  Arms: Gero-Erat

SUMMARY:
Currently, there is evidence that structured care within the healthcare system increases the conditions for good care and better recovery. We want to investigate whether a new care concept (gero-ERAT) that combines two variants of structured care can improve the recovery of elderly patients affected by a physical trauma.

Our hope is that the project will reduce the complications, short care times, fewer re-admissions and that more patients can return to regular living, which reduces the suffering for the patient and his relatives. In addition to patient benefit, a successful outcome will also result in reduced costs for healthcare and society as a whole. The concept of care is based on an increased patient participation, which is in line with the values of the Västra Götaland region and the Sahlgrenska university hospital

Through the PhD project, four studies will be published. A qualitative interview study to investigate patients' experiences of care and recovery after trauma.

After that, a prospective cohort survey of two groups is carried out; conventional care and gero-ERAT. Data will begin to be collected in the control group and when the control group is full geroRATAT will be implemented in the care department and we then collect data in the intervention group.

Based on collected data, we will publish two additional studies one with a focus on health economics as well as one focusing on care time and recovery based on age and harvest estimation.

DETAILED DESCRIPTION:
At present, there is evidence that structured care within healthcare (CGA and ERAS) increases the conditions for good care and better recoveries after acute conditions, planned and unplanned surgery. However, there are gaps in knowledge regarding elderly patients who are cared for within the surgical context. In this project we want to investigate whether a new care concept that combines CGA and ERAS can improve care and recovery for elderly patients who have suffered a physical trauma. We call care concepts for Geriatric Enhanced Recovery After Trauma (gero-ERAT). The project will be implemented as a PhD project for a maximum of 8 years. In the doctoral project, a qualitative interview study is planned during the spring and autumn of 2019. The purpose is to investigate experiences of care and recovery in elderly patients who have been cared for physical trauma. The findings from that study can contribute with new knowledge to the gero-ERAT concept.

The overall purpose of the project is to develop, implement and evaluate a structured care with the aim of improving care and recovery in elderly patients affected by physical trauma.

Specific purposes

1. Investigate patients experience of the recovery process after trauma
2. Establish, implement and evaluate the gero-ERAT concept (ie the effect of the intervention during the care period) at the trauma care unit at the university hospital.
3. Examine health economics when introducing and using gero-ERAT in the continuum care at the university hospital
4. Investigate in hospital time and recovery based on age and harvest estimation when using gero-ERAT

The first study will be a qualitative interview study, 20-25 (depending on when saturation of data occurs) patients will be deeply interviewed at approximately one hour.

The interviews will be semi-structured, and the questions are designed so that patients are given the opportunity to tell about their own perception and experience of care and recovery in connection with trauma. Transcribed coded data will be analyzed with the Constructive Grounded Theory methodology of Charmaz.

Potential participants will be asked by researchers who are involved in the project upon discharge from the hospital, patients receive both oral and written information. The patients will be interviewed approximately six weeks after discharge from the hospital and the interview session is expected to take between 1-3 hours.

The second study which is a Prospective cohort of two groups; conventional care and gero-ERAT will generate three studies.

Data will be collected from the patients journal and by surveys that the patient replies to The measurement variables will be collected in connection with the care period when the patient is included in the study (baseline value), as well as at six and 12 months after the patients have been written out from the hospital. The items 1-5 below will be collected via the patients' records and items 6-11 will be filled in by the patients.

* Demographic data (age, gender, type of trauma, other morbidity, social status, housing type)
* Length of stay
* Complications
* Re-admissions
* Mortality
* RAND-SF36 (Short Form Health Survey); is a validated generic questionnaire on health-related quality of life and consists of 36 questions that can be divided into two domains; physical and mental health.
* EQ-5D-5L (EuroQol); is a validated generic questionnaire consisting of five questions (health domains) and a VAS scale. In addition to health outcomes, data can be used as a basis for health economic calculations
* ADL (Activities in daily life) The staircase describes the degree of dependence / independence with three scale steps for five basic physical activities and a function (food intake, continence, movement, toilet visits, dressing and undressing and bathing).
* ESAS (Edmonton Symptom Assessment Scale); are validated symptom estimation scales consisting of ten symptoms (eg, pain, indigestion, nausea).
* PREM (Patient Reported Experienced Measures) is a measure for measuring the patient's experience and satisfaction of care.
* The PRP Questionnaire (Post Operational Recovery Profile) is a validated form consisting of 19 questions regarding symptoms such as appetite, insomnia and concentration ability that can be answered with four options.

Descriptive data will be used to describe the groups. The differences between the groups will be calculated with Fisher's exact test for nominal data, Chi two test (X2) test for ordinal distribution, and normal distributed continuous variables will be calculated with Student t test or if continuous data is not normally distributed with Mann-Whitney U- Test.'

3. The third study will be a health-economic analysis that is based on data from the EQ-5D, which can be used to obtain quality-of-life weights to calculate quality-adjusted life years (QALY). Length of hospital stay, complications and re-admissions will also be collected and reported systematically. While working on this sub study, in addition to statistics, a person within the clinic with expertise in health-economic calculations will also be involved.

4. The fourth study will be Examining length of hospital stay and recovery based on age and frailty estimation when using gero-ERAT. These sub-group analyzes will take place on all collected data described in sub-study II. Before the statistical analyzes begin, consultation with statisticians will take into account the problem of the mass significance's ability to adjust for this.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 65 years old
* In hospital due to physical trauma
* Able to speak and understand Swedish

Exclusion Criteria:

* Documented palliative care
* Cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2019-05-09 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay (LOS) | One year
  Length of hospital stay (LOS) in days

SECONDARY OUTCOMES:
SF-36 | One year
  The Short Form (36) Health Survey is a 36-item generic HRQoL questionnaire assessing eight domains: Physical function, Role-physical, Bodily pain, General health, Vitality, Social function, Role-emotional and Mental health. The first four domains reflect physical health and the last four mental health. A score is calculated for each domain on a scale from 0 (worst possible health state) to 100 (best possible health state)
Euro Quality of life - 5D | One year
  This is a standardized instrument for measure health outcome, it consists of a descriptive system and a VAS (Visual Analogue Scale). The descriptive system comprises five dimensions: Mobility, Self-care, Usual activities, Pain/Discomfort and Anxiety/Depression. Each dimension has 5 levels: No problems, Slight problems, Moderate problems, Severe problems and Extreme problems. Each domains can be calculated to a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale between 0-100 (100 = best imaginable health; 0 = worst imaginable health)
The Katz ADL (Activities of Daily Living Index) | One year
  Measures the individuals physical function, based on six activities: Feeding, Bathing, Dressing, Toileting, Continence and Transferring. Scoring: Each function can be answered with a yes/no for independence. The answers are then summarized and the result is compared with a list of seven steps between A to G, which indicates the alternative that best meets the assessed person's need for help.
  A = Independent of assistance in all six activities B = Dependent on assistance with one of the activities C = Dependent on bathing / showering assistance and one more activity D = Depending on assistance with bathing, dressing and undressing, toilet visits and additional activities E = Depending on assistance with bathing, dressing and undressing, toilet visits and another activity F = Depending on assistance with bathing, dressing and undressing, toilet visits, transfer and another activity G = Dependent on assistance with all activities.
ESAS (Edmonton Symptom Assessment Scale) | One year
  Measuring symptoms and illness. ESAS is a tool that estimate nine common symptoms for patients within palliative care: Pain, Tiredness, Drowsiness, Nausea, Appetite, Depression, Anxiety, Shortness of breath and Well-being. Each symptom are reported on a 10-grade scale ranges from no problem to worst possible problems.
PREM (Patient Reported Experienced Measures) | One year
  Patients satisfaction with provided care
Postoperative Recovery Profile (PRP) | One year
  This questionnaire is intended for self-assessment of general recovery after surgery. The questionnaire contains 19 items common after surgery, each item is estimated with a 4-degree verbal category scale from hard to none. The answers is coded and transformed in to a number and calculated on a scale from 0-19 on how well the person has recovered after surgery where <7 is not recovered at all and 19 is fully recovered.
Complications | One year
  Measuring rate of complications six months and one year after trauma
Mortality | One year
  Mortality measured six months and one year after trauma
Readmissions | One year
  Readmissions do to the trauma during one year after trauma

CONTACTS AND LOCATIONS:
Overall Officials: My Engström, PhD, Principal Investigator — Sahlgrenska University Hospital, Department of Surgery.
Locations (1):
- Sahlgrenska university hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No